CLINICAL TRIAL: NCT06272227
Title: Effect of Alfacalcidol on Muscle Function in Osteoporosis Patients; Double-blinded Randomized Controlled Trial
Brief Title: Effect of Alfacalcidol on Muscle Function in Osteoporosis Patients
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 4-2023-0986
Record Dates: First submitted 2024-02-14; First posted 2024-02-22 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Sarcopenia
MeSH Terms: conditions — Sarcopenia | interventions — alfacalcidol; Denosumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- alfacalcidol (Experimental): alfacalcidol plus denosumab
  Interventions: Drug: alfacalcidol; Drug: Denosumab
- placebo (Placebo Comparator): placebo + denosumab
  Interventions: Drug: placebo; Drug: Denosumab

INTERVENTIONS:
Drug: alfacalcidol — Subjects assigned to arm 1 take two doses of alfacalcidol once a day for a total of 52 weeks from the day after baseline visit 2 to the day before the end of the test (visit 4).
  Arms: alfacalcidol
Drug: placebo — Subjects assigned to arm 2 take two doses of placebo once a day for a total of 52 weeks from the day after baseline visit 2 to the day before the end of the test (visit 4).
  Arms: placebo
Drug: Denosumab — denosumab

SUMMARY:
This study aims to investigate the potential improvement in muscle function, compared to the placebo group, through the concurrent administration of denosumab and alfacalcidol over a one-year period in postmenopausal women with functional sarcopenia and osteoporosis aged 65 and older. The study is planned as a double-blinded randomized controlled trial, intending to recruit a total of 340 participants. Primary outcome is the improvement in SPPB score of 0.5 or more compared to the control group.

DETAILED DESCRIPTION:
This trial is a double-blind, randomized phase 4 trial to evaluate whether alfacalcidol co-administration improves muscle function compared to the placebo group in functional sarcopenia women over 65 years of age who are taking denosumab for osteoporosis. This trial consists of four trial periods (Screening Visit 1, Baseline Visit 2, Visit 3 (26 weeks), and Visit 4 (52 weeks).

ELIGIBILITY:
Inclusion Criteria:

* 1) Females aged 65 and above. 2) Individuals with osteoporosis who are either currently on denosumab or planning to initiate denosumab treatment.

  3) Participants committed to a minimum of 1-year denosumab treatment. 4) Those who have not taken any active vitamin D supplements within 3 months prior to the baseline visit (Visit 2).

  5) Participants capable of walking. 6-1) Individuals with SPPB ≤ 9 meeting the criteria for low physical performance.

6-2) Individuals with SPPB scores of 10 or 11 and concurrently exhibiting low muscle strength (hand grip strength < 18kg) or gait speed < 1.0 m/s or chair stand test > 11s (sitting position) or a history of fractures (excluding skull, cervical spine, fingers, toes, and rib fractures) or a fall within the past year.

7) Individuals who have undergone DXA (Dual-energy X-ray Absorptiometry) within 6 months of the baseline visit (Visit 2).

8) Participants who, after receiving a detailed explanation of the clinical trial, have fully understood it, voluntarily decided to participate, and provided written consent to participate while agreeing to adhere to the precautions

Exclusion Criteria:

1. Individuals contraindicated for active vitamin D supplementation:

   * Patients with hypercalcemia or hyperphosphatemia. ② Those with a history of urolithiasis/nephrolithiasis.
2. Individuals contraindicated for denosumab treatment:

   ① Those planning or with unresolved invasive dental procedures such as extractions, dental implants, or oral surgery.
   * Individuals with hypoalbuminemia-corrected serum calcium outside the normal range.
3. Individuals with vitamin D deficiency, defined as a serum 25(OH)D concentration below 12 ng/mL (30 nmol/L).
4. Participants who have received continuous prednisolone (or equivalent glucocorticoid) at a dose of 5 mg or higher per day for at least 90 days within 6 months of the screening visit (Visit 1).
5. Individuals with severe malnutrition, indicated by a serum albumin level of 3.0 mg/dL or below.
6. Those in an acute immobility state due to reasons such as fracture, hospitalization, or surgery within 1 month of the baseline visit (Visit 2).
7. Individuals with severe underlying conditions:

   ① Patients with metastatic cancer.

   ② Those with severe renal impairment (estimated Glomerular Filtration Rate; eGFR) less than 15 mL/min/1.73m² or undergoing dialysis.

   ③ Individuals receiving oxygen therapy due to chronic obstructive pulmonary disease (COPD).

   ④ Those with decompensated liver cirrhosis and severe liver disease with complications due to portal hypertension
8. Individuals with physical limitations due to specific conditions other than muscle decline: ① Those incapable of communication, including severe dementia. ② Individuals undergoing drug therapy for neuro-muscular disorders such as Parkinson's disease or severe myasthenia.
9. Individuals with an SPPB score of 12, indicating no impairment in physical function

Min Age: 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 340 (Estimated)
Dates: Start 2024-02-13 (Estimated); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Improvement in SPPB score of 0.5 or more compared to the control group | one year
  Our study aim is to demonstrate the improvement in SPPB(Short physical performace battery) score of 0.5 or more in the alfacalcidol group compared to the placebo group.

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Endocrinology, Department of internal Medicine, Yonsei University College of Medicine, Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No